CLINICAL TRIAL: NCT00196846
Title: Prospective Randomized Multicenter Study to Prevent Chemotherapy Induced Ovarian Failure With the GnRH-Agonist Goserelin in Young Hormone Insensitive Breast Cancer Patients Receiving Anthracycline Containing (Neo-)Adjuvant Chemotherapy
Brief Title: Prevention of Chemotherapy Induced Ovarian Failure With Goserelin in BC Patients (ZORO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Responsible Party: Konstantin Reißmüller, GBG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GBG37; Eudract Number: 2004-003980-62
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Breast Cancer
Keywords: hormone insensitive breast cancer; Prevention of Chemotherapy induced ovarian failure; P.O.F.; GnRH-Agonist Goserelin
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Goserelin

SUMMARY:
Study done in young breast cancer patients to prevent chemotherapy induced ovarian failure

DETAILED DESCRIPTION:
Study Design:

Prospective, randomized, open phase II trial

Schedule:

All patients will receive an anthracycline-containing polychemotherapy.

Patients randomized to Goserelin will receive their first injection of 3.6 mg at least 2 weeks before start of chemotherapy. Goserelin will be given as a subcutaneous injection in the abdominal wall every 4 weeks (28 ± 3 days) until the end of the last chemotherapy cycle.

Primary objective:

•To increase the percentage of patients with normal ovarian function at 6 months after application of (neo)adjuvant, anthracycline-containing polychemotherapy in parallel with Goserelin compared to chemotherapy alone.

Secondary objectives:

To compare the two treatment groups regarding

* Compliance to treatment
* Toxicity
* Quality of life
* Menopausal Symptoms Score
* Ovarian function at 6, 12, 18 and 24 months
* Duration until recovery of regular menstrual period
* Pregnancy rate

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained and documented according to the local regulatory requirements prior to beginning specific protocol procedures
* Complete baseline documentation sent to GBG
* Age of at least 18 and at most 45 years
* Patients request to preserve ovarian function
* Spontaneous and regular menstrual periods before study entry with FSH below 15 mlU/ml in follicular phase
* Histologically confirmed primary breast cancer with the need for anthracycline-based chemotherapy
* Steroid receptor (estrogen and progesterone) negative tumor (diagnosis according to hospital standard-procedures)
* No clinical evidence of local recurrence or distant metastases. Complete staging work-up within 3 months prior to registration. All patients must have (bilateral) mammography or breast MRI, chest X-ray; other tests may be performed as clinically indicated
* Karnofsky-Index >80%
* Life expectancy of at least 10 years, disregarding the diagnosis of cancer
* Adequate organ function including normal red and white blood count, platelets, serum creatinine, bilirubin, and transaminases within normal range of the institution
* Patients must be available for and compliant to treatment and follow-up. Patients registered on this trial must be treated and followed up at the participating center.

Exclusion Criteria:

* Known hypersensitivity reaction to the investigational compounds or incorporated substances
* Prior cytotoxic treatment for any reason
* Suspected (primary or secondary) ovarian insufficiency
* Pregnant or lactating patients. Patients of childbearing potential must have a negative pregnancy test (urine or serum) within 14 days prior to registration and must implement adequate non-hormonal contraceptive measures during study treatment; prior use of hormonal contraceptives has to be discontinued before first Goserelin injection
* Other serious illness or medical condition that may interfere with the understanding and giving of informed consent and the conduct of the study
* Prior or concomitant secondary malignancy (except non-melanomatous skin cancer or carcinoma in situ of the uterine cervix)
* Concurrent treatment with other experimental drugs or any other anti-cancer therapy
* Concurrent treatment with sex hormones. Prior treatment must be stopped before study entry

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2005-03; Primary Completion 2008-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Normal ovarian function as defined by two consecutive menstrual periods within 21-35 days within a time frame of 5 - 8 months after last application of goserelin | December 2008

SECONDARY OUTCOMES:
Discontinuation, delay, or dose-reductions of chemotherapy | December 2008
Discontinuation or delay of Goserelin injections | December 2008
Any grade II to grade IV AE specified to serious or non serious events during treatment with chemotherapy +/- Goserelin | December 2008
Evaluation according to EORTC Q 30 | March 2010
According to menopausal symptom score: E2, FSH, LH, SHGB, and Progesterone at 0, 6, 12, 18 and 24 months | March 2010
Date of first regular menstrual period | March 2010
Any diagnosis of pregnancy during study follow up | March 2010

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Gerber, MD, Principal Investigator — Rostock Universität, Universitätsfrauenklinik
Locations (1):
- Universitätsfrauenklinik, Rostock Universität, Rostock, Mecklenburg-Vorpommern, Germany

REFERENCES:
- See also: Click here for more information about this study: ZORO Study — http://www.germanbreastgroup.de